CLINICAL TRIAL: NCT04886531
Title: An Open Label, Phase II Trial of Pre-operative Neratinib and Endocrine Therapy With Trastuzumab in ER-Positive, HER-2 Positive Cancers Hoosier Cancer Research Network BRE17-141
Brief Title: Trial of Pre-operative Neratinib and Endocrine Therapy With Trastuzumab in ER-Positive, HER-2 Positive Breast Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruth O'Regan (Other)
Collaborators: Puma Biotechnology, Inc. (Industry); University of Rochester (Other)
Responsible Party: Sponsor-Investigator, Ruth O'Regan, Sponsor Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN BRE17-141
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer; ER Positive Breast Cancer; PR-Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Letrozole; Anastrozole; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- A (Experimental): Weeks 1-3* patients receive either (a) Neratinib, (b) Letrozole or Anastrozole or (c) Neratinib + Letrozole or Anastrozole
  Weeks 4-24 patients receive Neratinib + Letrozole or Anastrozole and Trastuzumab
  *Starting drug intervention varies for the first 3 weeks depending on arms: a, b, and c by randomization.
  Interventions: Drug: Neratinib; Drug: Letrozole (L) or Anastrozole (A); Drug: Trastuzumab

INTERVENTIONS:
Drug: Neratinib — 120mg for 7 days; 160mg for 7 days ; 240mg for 7 days. 240 mg (up to a maximum of 24 weeks) orally daily*.
  Other Names: Nerlynx
Drug: Letrozole (L) or Anastrozole (A) — L: (2.5 mg) OR A: (1 mg) orally daily (up to a maximum of 24 weeks)*
  Other Names: Femara; Arimidex
Drug: Trastuzumab — All Arms 8mg/kg loading dose followed by 6mg/kg every 3 weeks administered every 3 weeks by IV starting wk 4. Trastuzumab biosimilars may be used per institutional guidelines.
  Other Names: Herceptin

SUMMARY:
Patient will be treated with neratinib, an aromatase inhibitor and trastuzumab for 24 weeks prior to surgery, following an initial 3 weeks of neratinib alone, aromatase inhibitor alone or the combination of neratinib and an aromatase inhibitor. A breast biopsy will be performed prior to Day 1 of week 4 of treatment. Following surgery, patients will receive standard of care HER2-directed and endocrine therapy at the treating physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* Postmenopausal females. NOTE: Postmenopausal status defined as: prior bilateral oophorectomy, Age ≥ 60 years, or Age < 60 years and amenorrhea for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression) or an estradiol level in postmenopausal ranges per local reference range.
* ECOG Performance Status of 0-2 within 28 days prior to registration.
* Anatomic, clinical stage I-III, invasive breast cancer, greater than 10mm
* HER2-positive (by the most recent ASCO-CAP criteria)
* ER positive (≥ 10%). NOTE: There is no requirement for PR status; PR positive or negative allowed.
* Resectable breast cancer in which pre-operative therapy is appropriate (T > 10mm and/or node-positive).
* Archival tissue from the diagnostic pre-treatment biopsy is required. This sample should be identified at screening and shipped by Week 4. If archival tissue is not available, the subject is not eligible for the study.
* Agreeable to repeat breast biopsy at 3 weeks after initiation of treatment.
* Candidate for either letrozole or anastrozole, as determined by the treating physician
* Left ventricular ejection fraction (LVEF) ≥ 50% as assessed by echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) documented within 4 weeks prior to the study treatment.
* Demonstrate adequate organ function as defined below; all screening labs to be obtained within 28 days prior to registration.

  * Hematological

    * Platelet count ≥100,000/uL
    * Absolute Neutrophil Count (ANC) ≥1500/uL
    * Hemoglobin (Hgb) ≥10 g/dL
  * Renal

    ---Calculated creatinine clearance: CrCl ≥30 mL/min using the Cockcroft-Gault formula
  * Hepatic

    * Bilirubin ≤1.5 x upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) ≤ 2.5 × ULN
    * Alanine aminotransferase (ALT) ≤ 2.5 × ULN
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial.
* For patients with known serologic evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial.
* Ability of the subject to understand and comply with study procedures for the entire length of the study, as determined by the enrolling physician or protocol designee.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Locally advanced or inflammatory breast cancer. NOTE: Locally advanced is defined as Stage IIIC or greater.
* Evidence of metastatic disease. Systemic imaging is not required.
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are not eligible for this trial: exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
* Active infection requiring systemic therapy.
* Requirement for use of a moderate or strong CYP3A4 inhibitor or inducer during the study (see protocol).
* Treatment with any investigational drug within 14 days prior to registration or within 5 half-lives of the investigational product, whichever is longer.
* Subject has had major surgery within 14 days prior to registration or has not recovered from major side effects of the surgery (tumor biopsy is not considered as major surgery).
* Any impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection) or significantly impair the ability to swallow capsules/tablets.
* Known history of myelodysplastic syndrome or acute myeloid leukemia.
* Subjects with any of the following conditions:

  * History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 28 days prior to registration.
  * Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to registration.
  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to registration.
  * Symptomatic congestive heart failure (New York Heart Association III-IV) or documented current cardiomyopathy with left ventricular ejection fraction (LVEF) <50%.
  * Clinically significant cardiac ventricular arrhythmias (e.g. sustained ventricular tachycardia/ventricular fibrillation) or high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block) unless a pacemaker is in place.
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome.
* Any concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate subject participation in the clinical study or compromise compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | 24 weeks
  pCR is defined as the lack of all signs of invasive cancer in the breast removed during surgery

SECONDARY OUTCOMES:
Assess Adverse Events | 24 weeks
  Assess the adverse events of neratinib in combination with NSAI in subjects
Pathological Complete Response (pCR) | 24 weeks
  Estimate the pCR (ypT0/Tis ypN0) in the breast tissue and lymph nodes
Measure Residual Disease | 24 weeks
  Estimate residual disease in the breast tissue

CONTACTS AND LOCATIONS:
Overall Officials: Ruth O'Regan, MD, Principal Investigator — University of Rochester
Locations (4):
- United States (4):
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Rochester Medical Center, Rochester, New York
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No